CLINICAL TRIAL: NCT00395733
Title: A Single-blind, Intra-individual, Crossover, Multicenter Study of the Efficacy, Safety and Tolerability of Gadavist (1.0 M) in Comparison With Magnevist (0.5 M) as Contrast Agent in the Enhanced Magnetic Resonance Angiography (MRA) in Chinese Patients
Brief Title: Efficacy and Safety Study to Evaluate Gadavist (Gadobutrol) as Contrast Agent in Magnetic Resonance Imaging (MRI) of Vascular Diseases in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 91537; 309762 (Other: Company internal)
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-11

CONDITIONS: Vascular Diseases
Keywords: Gadovist; Gadavist; MRI Imaging; vascular diseases; Chinese
MeSH Terms: conditions — Vascular Diseases | interventions — gadobutrol; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gadobutrol, then Gadopentate dimeglumine (Experimental): Period 1: Participant received Gadobutrol 1.0 M (iv: intravenous injection), at a dose of 0.2 mL/kg BW, up to 0.3 mL/kg BW if 3 Fields of View (FOVs) to be imaged; Period 2: Participant received Gadopentate 0.5 M (iv), at a dose of 0.4 mL/kg BW, up to 0.6 mL/kg BW if 3 FOVs to be imaged
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875); Drug: Gadopentate dimeglumine (Magnevist, BAY86-4882)
- Gadopentate, dimeglumine then Gadobutrol (Experimental): Period 1: Participant received Gadopentate 0.5 M (iv), at a dose of 0.4 mL/kg BW, up to 0.6 mL/kg BW if 3 FOVs to be imaged; Period 2: Participant received Gadobutrol 1.0 M (iv: intravenous injection), at a dose of 0.2 mL/kg BW, up to 0.3 mL/kg BW if 3 Fields of View (FOVs) to be imaged
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875); Drug: Gadopentate dimeglumine (Magnevist, BAY86-4882)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW)
Drug: Gadopentate dimeglumine (Magnevist, BAY86-4882) — Participant received a single intravenous injection with Gadopentate (0.5 M) at a volume of 0.4 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.6 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW)

SUMMARY:
The purpose of this study is to determine if the contrast agent is effective and safe in the Magnetic Resonance Imaging (MRI) of vascular diseases in patients of Chinese origin.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* Known or suspected blood vessel diseases

Exclusion Criteria:

* Pregnancy
* Lactation
* Conditions interfering with MRI
* Allergy to any contrast agent or any drugs
* Participation in other trial
* Require emergency treatment
* Severely impaired liver and kidney functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- China (3):
  - Chengdu, Sichuan
  - Beijing
  - Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at specialized study centers if they satisfied the inclusion and exclusion criteria. All had known or suspected stenosis of arterial vessels in different vascular body regions with an indication for contrast-enhanced magnetic resonance angiography for diagnosis and further treatment.
Pre-assignment Details: Of 87 screened participants, 4 were not randomized (2 due to withdrawal of consent, 1 due to entering another clinical study and 1 was lost to follow-up). Thus, 83 participants were randomized to either the sequence Gadobutrol/Gadopentate dimeglumine (41 participants) or Gadopentate dimeglumine/Gadobutrol (42 participants).
Groups:
- Period 1: Gadobutrol, Period 2: Gadopentate Dimeglumine: Period 1: Gadobutrol 0.2 - 0.3 mmol/kg Body Weight (BW) (Gadavist, BAY86-4875); Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW). Period 2: Gadopentate dimeglumine 0.2 - 0.3 mmol/kg BW (Magnevist, BAY86-4882); Participant received a single intravenous injection with Gadopentate (0.5 M) at a volume of 0.4 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.6 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW).
- Period 1: Gadopentate Dimeglumine, Period 2: Gadobutrol: Period 1: Gadopentate dimeglumine 0.2 - 0.3 mmol/kg BW (Magnevist, BAY86-4882); Participant received a single intravenous injection with Gadopentate (0.5 M) at a volume of 0.4 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.6 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW). Period 2: Gadobutrol 0.2 - 0.3 mmol/kg BW (Gadavist, BAY86-4875); Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW).
Period: Period 1
Arm/Group | Period 1: Gadobutrol, Period 2: Gadopentate Dimeglumine | Period 1: Gadopentate Dimeglumine, Period 2: Gadobutrol
Started | 41 | 42
Completed | 41 | 42
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Period 1: Gadobutrol, Period 2: Gadopentate Dimeglumine | Period 1: Gadopentate Dimeglumine, Period 2: Gadobutrol
Started | 41 | 42
Completed | 39 | 37
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Technical problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Period 1: Gadobutrol, Period 2: Gadopentate Dimeglumine: Period 1: Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW). Period 2: Participant received a single intravenous injection with Gadopentate (0.5 M) at a volume of 0.4 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.6 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW).
- Period 1: Gadopentate Dimeglumine, Period 2: Gadobutrol: Period 1: Participant received a single intravenous injection with Gadopentate (0.5 M) at a volume of 0.4 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.6 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW). Period 2: Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW).
- Total: Total of all reporting groups
Arm/Group | Period 1: Gadobutrol, Period 2: Gadopentate Dimeglumine | Period 1: Gadopentate Dimeglumine, Period 2: Gadobutrol | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (14.26) | 55.3 (11.21) | 53.1 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Vessel Segments Visualized With Diagnostic Quality
Description: Each arterial segment visualized in magnetic resonance angiography (MRA) enhanced by Gadavist and Magnevist was characterized by the on-site investigators and by three independent blinded readers (reader 1, 2 and 3) according to a five-point scale (none/not assessable, poor, moderate, good, excellent), which takes into consideration intravascular contrast quality as well as vessel border delineation. The number of vessel segments with adequate diagnostic quality, i.e. good or excellent scores, was determined for each MRA image.
Time Frame: 20-30 seconds after injection
Population: Per Protocol Set (PPS): All participants who have received contrast injection and are not invalid cases. Note: The contrast enhanced MR image from one participant was lost after assessment by the investigator, i.e. the PPS analysis for the blinded readers is based on the images of 66 participants only.
Measure: Mean (Standard Deviation); unit: vessel segments
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Participant received a single intravenous injection with Gadobutrol (1.0 M) at a volume of 0.2 mL/kg BW (dose = 0.2 mmol/kg BW) or up to 0.3 mL/kg BW when 3 Fields of View were imaged (up to dose = 0.3 mmol/kg BW)
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 67 | 67
vessel segments
  Investigators | 8.10 (3.685) | 8.33 (3.755)
  Reader 1 | 8.03 (3.815) | 8.33 (3.852)
  Reader 2 | 7.55 (4.622) | 7.88 (3.665)
  Reader 3 | 5.27 (3.921) | 5.91 (3.666)
Statistical Analysis 1: Comparison: Gadobutrol (Gadavist, BAY86-4875) vs Gadopentate Dimeglumine (Magnevist, BAY86-4882); Non-inferiority analysis: The aim was to show that Gadavist is not inferior (i.e. similar or better) to Magnevist in visualizing different vascular regions of the body with diagnostic quality in contrast enhanced MRA. Gadavist was to be considered to be non-inferior to Magnevist if the mean number of vessel segments visualized with diagnostic quality of Gadavist enhanced-MRA images was higher than 85% of that of Magnevist enhanced-MRA images in a cross-over design; Test type: Non-Inferiority or Equivalence — Estimates for investigators only. A non-inferiority margin of 15% was assumed. Based on 60 pairs of observations in a crossover design (15 participants with 10 vessels segments, 15 participants with 6 vessels segments and 30 participants with 17 vessels segments to be visualized and assessed) and non-inferiority testing based the lower limit of Fieller's one-sided 95% confidence interval for the ratio Gadavist / Magnevist of the means, the power was at least 80% under realistic assumptions; Fieller-type confidence interval; Ratio of means = 0.9736, 90% CI [0.9315 to 1.0168] — For the estimation, only vessel segments with vascular assessments available for both periods were considered. The lower limit of the 95% one-sided Fieller-type confidence interval was compared with the non-inferiority margin 0.85
Statistical Analysis 2: Comparison: Gadobutrol (Gadavist, BAY86-4875) vs Gadopentate Dimeglumine (Magnevist, BAY86-4882); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Estimates for blinded reader 1 only. A non-inferiority margin of 15% was assumed. Based on 60 pairs of observations in a crossover design (15 participants with 10 vessels segments, 15 participants with 6 vessels segments and 30 participants with 17 vessels segments to be visualized and assessed) and non-inferiority testing based the lower limit of Fieller's one-sided 95% confidence interval for the ratio Gadavist / Magnevist of the means, the power was at least 80% under realistic assumptions; Fieller-type confidence interval; Ratio of means = 0.9540, 90% CI [0.9122 to 0.9965] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Gadobutrol (Gadavist, BAY86-4875) vs Gadopentate Dimeglumine (Magnevist, BAY86-4882); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Estimates for blinded reader 2 only. A non-inferiority margin of 15% was assumed. Based on 60 pairs of observations in a crossover design (15 participants with 10 vessels segments, 15 participants with 6 vessels segments and 30 participants with 17 vessels segments to be visualized and assessed) and non-inferiority testing based the lower limit of Fieller's one-sided 95% confidence interval for the ratio Gadavist / Magnevist of the means, the power was at least 80% under realistic assumptions; Fieller-type confidence interval; Ratio of means = 0.9458, 90% CI [0.8776 to 1.0240] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Gadobutrol (Gadavist, BAY86-4875) vs Gadopentate Dimeglumine (Magnevist, BAY86-4882); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Estimates for blinded reader 3 only. A non-inferiority margin of 15% was assumed. Based on 60 pairs of observations in a crossover design (15 participants with 10 vessels segments, 15 participants with 6 vessels segments and 30 participants with 17 vessels segments to be visualized and assessed) and non-inferiority testing based the lower limit of Fieller's one-sided 95% confidence interval for the ratio Gadavist / Magnevist of the means, the power was at least 80% under realistic assumptions; Fieller-type confidence interval; Ratio of means = 0.8698, 90% CI [0.7800 to 0.9657] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Diagnostic Confidence From Pre- to Post-contrast MRA by Investigator
Description: The on-site investigators assessed the change in diagnostic confidence in the assessment of MRA scans before and after injection with Gadavist and Magnevist for each participant on a three-point scale as improved, unchanged or worsened.
Time Frame: immediately before and 20-30 seconds after injection (precontrast and postcontrast)
Population: Per Protocol Set (PPS): All participants who have received contrast injection and are not invalid cases.
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 67 | 67
Participants
  improved | 63 | 65
  unchanged | 0 | 0
  worsened | 0 | 0
  missing or not applicable | 4 | 2

3. Secondary Outcome: Change in Diagnostic Confidence From Pre- to Post-contrast MRA by Blinded Reader 1
Description: Independent blinded reader 1 assessed the change in diagnostic confidence in the assessment of MRA scans before and after injection with Gadavist and Magnevist for each participant on a three-point scale as improved, unchanged or worsened.
Time Frame: immediately before and 20-30 seconds after injection (precontrast and postcontrast)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Participants
  improved | 61 | 63
  unchanged | 0 | 0
  worsened | 1 | 0
  missing or not applicable | 4 | 3

4. Secondary Outcome: Change in Diagnostic Confidence From Pre- to Post-contrast MRA by Blinded Reader 2
Description: Independent blinded reader 2 assessed the change in diagnostic confidence in the assessment of MRA scans before and after injection with Gadavist and Magnevist for each participant on a three-point scale as improved, unchanged or worsened.
Time Frame: immediately before and 20-30 seconds after injection (precontrast and postcontrast)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Participants
  improved | 56 | 63
  unchanged | 3 | 1
  worsened | 1 | 0
  missing or not applicable | 6 | 2

5. Secondary Outcome: Change in Diagnostic Confidence From Pre- to Post-contrast MRA by Blinded Reader 3
Description: Independent blinded reader 3 assessed the change in diagnostic confidence in the assessment of MRA scans before and after injection with Gadavist and Magnevist for each participant on a three-point scale as improved, unchanged or worsened.
Time Frame: immediately before and 20-30 seconds after injection (precontrast and postcontrast)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Participants
  improved | 59 | 63
  unchanged | 0 | 0
  worsened | 2 | 0
  missing or not applicable | 5 | 3

6. Secondary Outcome: MRA Diagnosis by Investigators
Description: The MRA diagnosis describes the pathology with regard to the extent of a stenosis, i.e., normal (no relevant disease), advanced arteriosclerosis but stenosis <= 50% (exemption: internal carotid artery: stenosis <= 70%), advanced arteriosclerosis, stenosis >50% but <99% (stenosis 50-99%) (exemption: internal carotid artery >70%), occlusion, and not assessable.
Time Frame: 20-30 seconds after injection
Population: Per Protocol Set (PPS): All participants who have received contrast injection and are not invalid cases.
Measure: Number; unit: Vessels
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 67 | 67
Vessels
  100% diameter reduction (occlusion) | 6 | 8
  normal | 494 | 504
  <= 50% stenosis | 47 | 30
  > 50% stenosis | 32 | 32
  stenosis <= 70% | 5 | 3
  stenosis > 70% | 0 | 0
  not assessable | 271 | 278

7. Secondary Outcome: MRA Diagnosis by Blinded Reader 1
Description: as for outcome 6
Time Frame: 20-30 seconds after injection
Population: as for outcome 1
Measure: Number; unit: Vessels
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Vessels
  100% diameter reduction (occlusion) | 5 | 5
  normal | 503 | 497
  stenosis <= 50% | 33 | 37
  stenosis > 50% | 22 | 24
  stenosis <= 70% | 2 | 1
  stenosis > 70% | 1 | 1
  not assessable | 272 | 273

8. Secondary Outcome: MRA Diagnosis by Blinded Reader 2
Description: as for outcome 6
Time Frame: 20-30 seconds after injection
Population: as for outcome 1
Measure: Number; unit: Vessels
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Vessels
  100% diameter reduction (occlusion) | 15 | 10
  normal | 503 | 549
  <= 50% stenosis | 83 | 38
  > 50% stenosis | 21 | 16
  stenosis <= 70% | 1 | 1
  stenosis > 70% | 0 | 0
  not assessable | 215 | 224

9. Secondary Outcome: MRA Diagnosis by Blinded Reader 3
Description: as for outcome 6
Time Frame: 20-30 seconds after injection
Population: as for outcome 1
Measure: Number; unit: Vessels
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66 | 66
Vessels
  100% diameter reduction (occlusion) | 3 | 2
  normal | 489 | 499
  <= 50% stenosis | 8 | 11
  > 50% stenosis | 15 | 17
  stenosis <= 70% | 2 | 1
  stenosis > 70% | 0 | 0
  not assessable | 321 | 308

ADVERSE EVENTS:
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) | Gadopentate Dimeglumine (Magnevist, BAY86-4882)
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/81
Other Adverse Events (participants affected / at risk) | 7/78 | 7/81
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=78) | Gadopentate Dimeglumine (Magnevist, BAY86-4882) (N=81)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs shall provide sponsor with an advance copy of any proposed publication or oral presentation at least ninety (90) days prior to the date of the planned submission or presentation. Sponsor shall have sixty (60) days to recommend any changes it reasonably believes are necessary for scientific purposes or to preserve the confidentiality of sponsor's confidential information. PIs agree that the adoption of such recommended changes shall not be unreasonably refused.